CLINICAL TRIAL: NCT00786916
Title: Efficacy of Intravenous Lidocaine at Alleviating Pain Associated With Propofol Infusion in Pediatric Patients Undergoing Procedural Sedation
Brief Title: Efficacy of IV Lidocaine at Alleviating Pain Associated With Propofol Infusion in Pediatric Patients Undergoing Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael D. Reed, Pharm.D., Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 080209
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: pain; propofol; lidocaine; sedation; pediatric
MeSH Terms: conditions — Pain | interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Placebo Comparator): Saline
  Interventions: Drug: normal saline
- Group B (Active Comparator): Lidocaine 0.25 mg/kg
  Interventions: Drug: lidocaine
- Group C (Active Comparator): Lidocaine 0.5 mg/kg
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: normal saline — A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive saline placebo IV (Group A) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
  Arms: Group A
Drug: lidocaine — A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive lidocaine 0.25 mg/kg IV (Group B) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
  Arms: Group B
Drug: lidocaine — A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive lidocaine 0.5 mg/kg IV (Group C) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
  Arms: Group C

SUMMARY:
This protocol describes a double-blind, placebo-controlled trial intended to demonstrate the effectiveness of lidocaine at reducing pain associated wiht propofol infusion for short-term deep sedation in children. Patients will be randomized to receive either placebo (saline) or one of two dosing regimens of IV lidocaine prior to initiating propofol infusion. The efficacy of the differing lidocaine doses will be compared to determine the minimum dose required to safely achieve alleviation of pain. We hypothesize that premedicating with lidocaine will significantly decrease pain experienced by pediatric patients receiving propofol for outpatient sedation.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for painless diagnostic procedures
* are ASA I or ASA II

Exclusion Criteria:

* have an indwelling central venous catheter
* have received an analgesic or sedative medication in the previous four hours prior to enrollment
* have an underlying chronic disorder that would impact on their ability to express distress when in painful or otherwise anxiety-provoking situations
* known hypersensitivity to lidocaine or any component of the formulation
* hypersensitivity to another local anesthetic of the amide type
* Adam-Stokes syndrome
* severe degrees of SA, AV, or intraventricular heart block
* allergy to corn-related products
* contraindication to propofol

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman C Christopher, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized, double-blind study was conducted at Akron Children's Hospital. The enrollment period was from 4/8/2008 to 2/9/2010.
Pre-assignment Details: Patients between 2 and 7 years of age with ASA 1 or ASA 2 classification and scheduled for painless diagnostic procedures were eligible for exclusion.
Groups:
- Group A: Saline
  normal saline : A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive saline placebo IV (Group A) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
- Group B: Lidocaine 0.25 mg/kg
  lidocaine : A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive lidocaine 0.25 mg/kg IV (Group B) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
- Group C: Lidocaine 0.5 mg/kg
  lidocaine : A blood pressure cuff is placed with its distal-most margin 10 cm proximal to the intravenous catheter insertion site and is inflated to 40 mmHg of pressure greater than the patient's pre-procedure systolic blood pressure. Subjects will receive lidocaine 0.5 mg/kg IV (Group C) prior to initiating propofol infusion. Five minutes after administration of the study agent, tourniquet pressure is released and propofol infusion will be immediately initiated.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 39 | 36 | 34
Completed | 39 | 36 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 39 | 36 | 34 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 36 | 34 | 109
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.61) | 4.3 (1.50) | 5.0 (1.63) | 4.67 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 15 | 43
  Male | 26 | 21 | 19 | 66
Region of Enrollment [Number; unit: participants]
  United States | 39 | 36 | 34 | 109

OUTCOME MEASURES:

1. Primary Outcome: Maximal Pain/Discomfort
Description: FLACC (Face, Legs, Activity, Cry, Consolability) Pain assessment scale was administered by a trained observer. The patient's parent documented maximum distress using a 100-mm visual analog scale where "0" represented "no pain" and 100 (the furthest point to the left) represented the worst pain ever.
Time Frame: during initial 3 minute propofol infusion
Population: All enrolled subjects were randomized into groups A, B or C by hospital pharmacists utilizing a standard prerandomization methodology.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 39 | 36 | 34
units on a scale | 4.7 (1.61) | 4.3 (1.50) | 5.0 (1.63)

ADVERSE EVENTS:
Groups:
- Group A: Placebo (Saline) Group
- Group B: 0.25 mg/kg Lidocaine Group
- Group C: 0.50 mg/kg Lidocaine Group
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/39 | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
No complications or adverse reactions were associated with either study drug dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes